CLINICAL TRIAL: NCT01048957
Title: The Neural Basis of Cue-Elicited Cigarette Craving and Its Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Purpose: Other
Other Study IDs: 999907418; 07-DA-N418
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2013-04-08

CONDITIONS: Nicotine Dependence
Keywords: Nicotine; Craving; fMRI; EEG; Real Time fMRI Feedback
MeSH Terms: conditions — Tobacco Use Disorder

INTERVENTIONS:
Behavioral: Real Time Feedback Training

SUMMARY:
Background:

- One kind of drug craving, known as cue-elicited craving, occurs when a drug user who sees a drug-related cue (such as an image of someone using the drug) begins to feel a craving for the drug. Researchers are interested in studying how cue-elicited craving affects brain activity using functional magnetic resonance imaging (fMRI) and electroencephalography (EEG) data.

Objectives:

- To determine which parts of the brain are associated with or involved in controlling cue-related craving in smokers.

Eligibility:

- Individuals between 18 and 50 years of age who are current smokers (10 or more cigarettes per day) and agree to try to abstain from smoking for 1 week during the experiment.

Design:

* Participants will visit a clinical center for up to four scanning sessions, and will be asked to perform two or three outpatient tasks at home over the course of the study.
* Scan 1: Training session with a mock fMRI scanner, followed by an actual fMRI scanning session and EEG in which participants respond to pictures.
* Outpatient Task 1: Tolerance test with nicotine patch (worn for 8 hours, followed by 12 additional hours without cigarette use).
* Scans 2 and 3: Training session and fMRI scan and testing with either nicotine patch or placebo. Tasks in fMRI involve looking at cues, reporting craving and suppressing craving.
* Outpatient Task 2: Participants will keep an electronic diary for 10 to 14 days, responding to questions as directed by the researchers.
* Scans 4 and 5: Training session, fMRI scan and EEG, and testing in which participants will be instructed on methods to attempt to control cravings.
* Outpatient Task 3: Participants will keep an electronic diary for 14 days. For the first 7 days, participants will be asked to attempt to abstain from nicotine; participants may smoke normally on the second 7 days.
* Participants will be contacted 1, 3, 6, and 12 months after the end of the study for follow-up questions on current smoking habits.

DETAILED DESCRIPTION:
Objective: Drug craving is a motivational state associated with a conscious desire to consume a drug (Fredrickson et al., 1995; Drummond, 2001). When drug abusers see drug-related cues, cue-elicited drug craving is induced (Drummond, 2001). The main goal of this investigation is to ascertain the neural basis of cue-elicited drug (e.g. cigarette) craving and its control in smokers.

Study population: The experimental population for this investigation is nicotine-dependent adults aged 18-50 years old.

Design: Participants will see the smoking-related cue or neutral cue and complete cognitive tasks (e.g. to report or regulate their craving, etc). At same time, we will employ functional magnetic resonance imaging (fMRI), real-time functional magnetic resonance imaging (rtfMRI), and electroencephalography (EEG) to measure brain activity.

Outcome measures: There is no direct benefit to the participant by joining this study. Data from this study are expected to contribute to a better understanding of the neural processes of cigarette craving. Thus, the results may benefit the health of society. MRI-related risks (e.g., injury from metal implants, claustrophobia, and temporary hearing threshold alterations due to the loud banging noises) and nicotine-patch-related risks (e.g., dizziness, headache, upset stomach, vomiting, diarrhea, redness or swelling at the patch site) to participants are minimized by careful prescreening and standard protection.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants must:

1. Be between the ages of 18-50. Justification: Many cognitive processes change with age. In addition, the risk of difficult-to-detect medical abnormalities such as silent cerebral infarcts increases with age. Therefore, older individuals, defined as those over 50, will be excluded.
2. Be in good health. Justification: Many illnesses can alter fMRI signal, and cognition. Assessment tool(s): Participants will provide a brief health history during phone screening, and undergo a history and physical examination with a qualified IRP clinician.
3. Be right-handed. Justification: Many of the brain functions to be assessed in this protocol have shown some evidence of being lateralized in the brain. In order to reduce the variance in the data from this possibility, participants must be right-handed. Assessment tool(s): Edinburgh Handedness Inventory
4. Be free of dependence on other substances (except nicotine). Justification: Dependence on other substances may result in unique CNS deficits that would increase the noise in our data. Assessment tool(s): Substance Use Disorders module of the SCID with confirmation by clinical interview and negative urine drug screen.
5. Must smoke greater than or equal to 10 cigarettes per day for at least two years, with urine cotinine levels of at least 100ng/ml and score on the Fagerstrom Test for Nicotine Dependence (FTND) must be greater than or equal to 2. Justification: The aim is to study phenomena that are linked to nicotine dependence and that occur with regular and frequent smoking. Assessment tool(s): Self-report, a urine cotinine test (smokers will be defined as having cotinine levels greater than or equal to 100ng/mL), and FTND test.
6. All participants should be able to abstain from alcohol for 24 hours and no more than 1/2 cup of caffeine for 12 hours before each experiment session. Justification: Alcohol and caffeine may result in brain that influences our data. Assessment tool(s): Self-report and breathalyzer test.

EXCLUSION CRITERIA:

Participants will be excluded if they:

1. Are not suitable to undergo an fMRI experiment due to pregnancy, implanted metallic devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts), body morphology or claustrophobia. Justification: MR scanning is one of the primary measurement tools used in the protocol. Assessment tool(s): Prospective participants will fill out an MRI screening questionnaire and undergo an interview with an MR technologist. Pregnancy tests will be performed on all female participants of childbearing age before each experimental session. Questions concerning suitability for scanning will be referred to the MR Medical Safety Officer. Prospective participants will be questioned about symptoms of claustrophobia and placed in the mock scanner during their first visit to assess for possible difficulty tolerating the confinement of the scanner and for ability to fit into the scanner.
2. Have coagulopathies, history of, current superficial, or deep vein thrombosis, musculoskeletal abnormalities restricting an individual s ability to lie flat for extended periods of time. Justification: MR scanning sessions require participants to lie flat on their backs and remain perfectly still for approximately two hours. Therefore, conditions that would make that difficult (e.g. chronic back pain, significant scoliosis) or dangerous (e.g. familial hypercoagulability syndrome, history of thrombosis) will be exclusionary. Assessment tool(s): History and physical examination by a qualified IRP clinician, supplemented with a trial of lying in the mock scanner to assess comfort issues.
3. Have HIV or Syphilis. Justification: HIV and Syphilis can both have CNS sequelae, thus introducing unnecessary variability into the data. Assessment tool(s): HIV blood test and RPR+.
4. Have any neurological illnesses to include, but not limited to, seizure disorders, migraine (>2/yr or on prophylaxis), multiple sclerosis, movement disorders, or history of significant head trauma, CVA, CNS tumor. Justification: CNS diseases alter CNS function and, possibly, the neuronal-vascular coupling that forms the basis of the BOLD fMRI signal to be used in this study. Assessment tool(s): History and physical examination by a qualified IRP clinician, urine drug screening for anticonvulsants not disclosed by history. History of head trauma with loss of consciousness of more than 5 minutes or with post-concussive sequelae lasting more than two days, regardless of loss of consciousness, will be exclusionary.
5. Have other major medical illnesses likely to interfere with study results or safety of an individual during participation. Justification: Many illness not covered here may increase risk or alter important outcome measures. Assessment tool(s): History and physical examination by a qualified IRP clinician and CBC, urinalysis, NIDA chemistry panel (liver function tests, electrolytes, kidney function). The following individual laboratory results will independently disqualify individuals. The MRP will retain discretion to exclude at less extreme values, depending on the clinical presentation, and will make the final judgment on any questionable lab results

   * Hemoglobin < 10 g/dl
   * WBC < 2400/microl
   * LFTs > 3 times normal
   * HCG positive
   * Serum glucose > 200 mg/dl
   * Urine protein > 2 plus
   * Serum cholesterol level> 250 mg/dl.
6. Have any current major psychiatric disorders to include, but not limited to, mood, anxiety, psychotic disorders, or substance-induced psychiatric disorders. Justification: Psychiatric disorders involve the central neural system (CNS) and, therefore, can be expected to alter the fMRI measures being used in this study. Assessment tool(s): Computerized SCID-NP, ASRS (adult ADHD self-report scale) and DSM-IV (DSM-IV, APA, 1994) confirmed by clinician interview.
7. Regularly use any prescription, over-the-counter or herbal medication that may alter CNS function, cardiovascular function or neuronal-vascular coupling. Justification: Compounds that alter BOLD signal will alter the primary measure used in the study. Assessment tool(s): History and comprehensive urine drug screening to detect antidepressants, benzodiazepines, antipsychotics, anticonvulsants, barbiturates and other common medications and drugs of abuse.
8. Are cognitively impaired or learning disabled. Justification: Cognitive impairment and learning disabilities are associated with alterations in brain regions used to accomplish tasks, and, therefore, may introduce significant variably into the data. In addition, cognitive impairment may affect ability to give informed consent. Assessment tool(s): History of known learning disability or cognitive impairment. Vocabulary subtest of the WASI will be given. IQ estimate must be over 85 (corresponding to a vocabulary subtest score > 48). In cases of suspected non-verbal learning disability or mild verbal deficit, a full WASI may be given to obtain a more robust estimate of IQ.
9. Significant cardiovascular or cerebrovascular diseases. Justification: Such conditions can alter and distort BOLD and autonomic signals and increase the risks associated with nicotine patch use. Assessment tool(s): History and physical exam, including 12-lead ECG.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2007-01-09; Primary Completion 2013-04-08 (Actual); Study Completion 2013-04-08 (Actual)

PRIMARY OUTCOMES:
To ascertain the neural basis of cue-elicited drug (e.g. cigarette) craving and its control in smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Andreasen NC, Endicott J, Spitzer RL, Winokur G. The family history method using diagnostic criteria. Reliability and validity. Arch Gen Psychiatry. 1977 Oct;34(10):1229-35. doi: 10.1001/archpsyc.1977.01770220111013. PMID 911222
- [Background] Aron AR, Fletcher PC, Bullmore ET, Sahakian BJ, Robbins TW. Stop-signal inhibition disrupted by damage to right inferior frontal gyrus in humans. Nat Neurosci. 2003 Feb;6(2):115-6. doi: 10.1038/nn1003. No abstract available. PMID 12536210
- [Background] Babiloni F, Mattia D, Babiloni C, Astolfi L, Salinari S, Basilisco A, Rossini PM, Marciani MG, Cincotti F. Multimodal integration of EEG, MEG and fMRI data for the solution of the neuroimage puzzle. Magn Reson Imaging. 2004 Dec;22(10):1471-6. doi: 10.1016/j.mri.2004.10.007. PMID 15707796